CLINICAL TRIAL: NCT04491084
Title: FLT3 Ligand (CDX-301), CD40 Agonist Antibody (CDX-1140), and Stereotactic Radiotherapy Versus Standard Therapy for Advanced Non-small Cell Lung Cancer: A Phase I/II Randomized Trial
Brief Title: FLT3 Ligand, CD40 Agonist Antibody, and Stereotactic Radiotherapy
Acronym: FLT3
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11868
Record Dates: First submitted 2020-07-21; First posted 2020-07-29 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: CDX-301; CDX-1140
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — flt3 ligand protein

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label phase I/II study. Subjects will be randomized in a 1:1 ratio to receive FLT3 ligand (CDX-301), anti-CD40 antibody (CDX-1140) and SBRT (Arm 1) versus standard care (Arm 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FLT3 ligand (CDX-301), anti-CD40 antibody (CDX-1140), and SBRT (Experimental): Subjects on either study arm with limited disease will receive SBRT to all evident sites of active disease. Subjects on Arm 1 with extensive disease will initially receive SBRT to a single site of disease but may receive additional "cycles" of FLT3 ligand, anti-CD40 antibody, and SBRT at later time points.
  Interventions: Drug: FLT3 Ligand (CDX-301); Biological: anti-CD40 antibody (CDX-1140); Radiation: SBRT
- Standard care (Active Comparator): Subjects on either study arm with limited disease will receive SBRT to all evident sites of active disease.Subjects on Arm 2 with extensive disease are expected to receive some form of standard systemic therapy (e.g., docetaxel). Subjects on Arm 2 with limited disease may also receive standard systemic therapy following completion of SBRT to all sites of evident disease, at the discretion of the treating physicians.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Drug: FLT3 Ligand (CDX-301) — Fms-like tyrosine kinase 3 (FLT3) ligand is a potent hematopoietic growth factor that mobilizes stem cells and greatly increases the number of circulating dendritic cells (DCs) in blood and organs.
  Arms: FLT3 ligand (CDX-301), anti-CD40 antibody (CDX-1140), and SBRT
Biological: anti-CD40 antibody (CDX-1140) — CD40 is a key molecule in the regulation of immune responses whose activity can be modulated using antibodies. CD40 is a tumor necrosis factor receptor superfamily member expressed on antigen presenting cells, including dendritic cells, as well as a host of other cell types, including a wide range of tumor cells
  Arms: FLT3 ligand (CDX-301), anti-CD40 antibody (CDX-1140), and SBRT
Radiation: SBRT — For subjects on Arm 1, SBRT will be delivered concurrently with FLT3 ligand during Week 1 of study therapy. If only one lesion is being treated, SBRT should be completed during week 1 (e.g., with daily treatments for a 5-fraction course of treatments every other day for a 3-fraction course). In cases where multiple lesions are being treated with SBRT (Arm 1 or Arm 2) or if treatment is interrupted due to technical issues or intercurrent illness, SBRT may extend beyond Week 1.

SUMMARY:
The purpose of this study is to test a new way of treating the most common form of lung cancer. The investigators are testing a combination of radiotherapy with two new forms of immunotherapy. This study is testing the safety and effectiveness of this treatment approach as compared to standard treatment options.

DETAILED DESCRIPTION:
This is a randomized, open-label phase I/II study. Subjects will be randomized in a 1:1 ratio to receive FLT3 ligand (CDX-301), anti-CD40 antibody (CDX-1140) and SBRT (Arm 1) versus standard care (Arm 2). Subjects on either study arm with limited disease will receive SBRT to all evident sites of active disease. Subjects on Arm 1 with extensive disease will initially receive SBRT to a single site of disease but may receive additional "cycles" of FLT3 ligand (CDX-301) anti-CD40 antibody (CDX-1140), and SBRT at later time points. Subjects on Arm 2 with extensive disease are expected to receive some form of standard systemic therapy (e.g., docetaxel). Subjects on Arm 2 with limited disease may also receive standard systemic therapy following completion of SBRT to all sites of evident disease, at the discretion of the treating physicians. All subjects will be followed closely for treatment-related toxicities. Whole-body PET/CT and CT imaging will be performed prior to study entry, and restaging CT will be performed every 8 weeks thereafter.

In the phase I component of this study, subjects will be randomized between study arms until 6 subjects have been randomized to Arm 1. Study accrual will then be halted until 8 weeks after the last study subject begins treatment.

If the pre-specified safety criteria are achieved in the Phase I portion of this study, the study will proceed to phase II. The total sample size (Phase I and Phase II) will be 46 subjects. All 46 subjects will be included in efficacy analyses.

If the pre-specified safety criteria are not achieved in the Phase I portion of this study, the investigators and Celldex will review safety data from this trial as well as other trials using CDX-301 and CDX-1140 and determine if the experimental treatment regimen should be altered (e.g., by reducing the CDX-1140 dose). The study protocol would be amended accordingly, and Phase I component with the new treatment regimen would be added.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC, not classically deemed to be amenable to curative therapy based on disease extent at the time of diagnosis or disease progression after the initial diagnosis
* Age ≥ 18 years
* Prior treatment with at least two lines of systemic therapy for advanced NSCLC, including one line of platinum-based combination chemotherapy
* Treatment with concurrent chemotherapy and immunotherapy can count as two lines of therapy for the purposes of study eligibility.
* Radiological assessment within 21 days prior to study entry demonstrating measurable disease that includes at least one pulmonary or extrapulmonary lesion ≥ 1 cm in greatest dimension that would be amenable to SBRT and at least one measurable lesion that would be outside of the SBRT treatment fields
* ECOG performance status 0-2
* Both men and women enrolled in this trial must agree to use adequate birth control measures during the trial and for at least 90 days after last receipt of study therapy. Patients and/or partners who are surgically sterile or postmenopausal are exempt from this requirement.
* The following laboratory results, within 21 days prior to first study drug administration (Arm 1) or within 21 days prior to study registration (Arm 2):

Hemoglobin ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Serum creatinine ≤ 1.5 x ULN OR creatinine clearance (by Cockcroft-Gault formula) > 60 mL/min AST and ALT ≤ 2.5 x ULN Total bilirubin ≤ 2.0 x ULN (except patients with Gilbert's syndrome, who must have a total bilirubin ≤ 3.0 mg/dL)

-Negative SARS-CoV-2 (COVID-19) PCR test. COVID-19 testing may be repeated periodically based on institutional policies and must be repeated for any subject with unexplained signs (e.g., imaging findings, fever) or symptoms (e.g., anosmia) concerning for COVID-19 infection or with recent known exposure to COVID-19.

Exclusion Criteria:

* Prior therapy with any anti-CD40 antibody or FLT3 ligand
* Less than 21 days between registration and the last receipt of chemotherapy, targeted cancer therapy, immunotherapy, radiotherapy (excluding palliative radiotherapy), or major surgery.
* Untreated central nervous system metastases. Patients with a history of brain metastases must have had no CNS-directed therapy within the past 60 days and radiological assessment within 30 days of study entry demonstrating a lack of progressive CNS disease. -Patients without a history of brain metastases and without symptoms suggestive of brain metastasis do not require staging imaging of the brain prior to study enrollment.
* Known mutation/amplification in FLT3
* Ongoing or recent (within 21 days prior to study entry) use of high dose oral corticosteroids (≥ 2 mg of dexamethasone daily or equivalent) or inhaled corticosteroids. Intranasal and/or intraarticular corticosteroid use is permitted.
* History of non-infectious pneumonitis or any ongoing pneumonitis
* History of allogeneic organ transplant or active autoimmune disease
* Other active malignancy for which systemic therapy (excluding hormonal therapy for breast or prostate cancer) is indicated.
* History of myocardial infarction, cerebral vascular accident, thrombosis, or pulmonary embolus within 12 months prior to study registration.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements as judged by the treating physicians
* Active infection requiring systemic therapy, known HIV infection, or positive test for hepatitis B surface antigen or hepatitis C (antibody screen and if positive confirmed by RNA analysis). If positive results are not indicative of a true active or chronic infection, the patient can be enrolled after discussion with, and agreement by, the Principal Investigator.
* Receipt of a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Subjects who are not ambulatory or ambulate using a walker are not eligible for the objective activity monitoring component of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 1 | 2
  Spanish/Hispanic/Latino | 0 | 2 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Dose-limiting Toxicity (DLT), Defined as Follows:
Description: Death
  Any ≥ Grade 3 non-hematological toxicity, with the following exceptions:
  Grade 3 alopecia, vitiligo, or endocrinopathies controlled by hormone replacement therapy Grade 3 nausea that resolves to ≤ grade 2 with or without treatment within 72 hours Grade 3 vomiting and diarrhea that resolves to ≤ grade 2 with or without treatment within 72 hours Grade 3 fatigue that resolves to ≤ grade 2 within 5 days Grade 3 hypertension in the absence of maximal medical therapy Grade 3 adverse event of tumor flare (defined as local pain, irritation, or rash localized at sites of known or suspected tumor) of ≤ 7 days in duration Grade 3 amylase or lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis. It is recommended to consult with the Principal Investigator for grade 4 amylase or lipase abnormalities
  Grade 3 clinically significant laboratory abnormalities that are asymptomatic and can be reversed within 72 hours, however:
  Any Grade 4
Time Frame: up to 8 weeks after initiation of study therapy
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Phase II: Progression-free Survival (PFS) Duration
Time Frame: defined as time from study registration until disease progression (scored using iRECIST) or death, whichever comes first up to 51 weeks.
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS) Duration
Description: Length of time that patient survives from time of study registration
Time Frame: From date of registration until the date of death from any cause, assessed up to 2 years
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Radiographic Responses Using Descriptive Statistics
Description: The clinical benefit rate (CBR) will be defined as the percentage of subjects who achieve best response of confirmed CR or PR, or stable disease (SD) for at least four months.
Time Frame: From date of registration, assessed up to 4 months
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life Using EORTC QLQ-LC13 (Quality of Life Questionnaire, Lung Cancer)
Description: Summary statistics (mean, standard deviation, median, 25th and 75th percentiles, and range) and the mean change from baseline of linear-transformed scores will be reported for all the items and subscales of the EORTC QLQ-C30 questionnaire and the QLQ-LC13, according to the EORTC scoring manual guidelines. higher scores are a better level of functioning
Time Frame: 1 year
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life Using QLQ-C30 (Quality of Life Questionnaire)
Description: Summary statistics (mean, standard deviation, median, 25th and 75th percentiles, and range) and the mean change from baseline of linear-transformed scores will be reported for all the items and subscales of the EORTC QLQ-C30 questionnaire and the QLQ-LC13, according to the EORTC scoring manual guidelines. Most items are scored 1 to 4, higher scores are a better level of functioning.
Time Frame: 1 year
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Daily Step Count Using Descriptive Statistics
Description: Average daily step counts
Time Frame: 1 year
Population: Data was not collected/aggregated. No analyses conducted.
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All participants enrolled in the trial were assessed through 49 weeks
Arm/Group | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT (N=2) | Standard Care (N=3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — Septic Shock
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hypoxic Respiratory Failure
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Recurrent hip pain leading to hospitalization
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) — Pneumonia
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Fall
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0) — Muscle weakness left-sided
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) — Dysarthria
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLT3 Ligand (CDX-301), Anti-CD40 Antibody (CDX-1140), and SBRT (N=2) | Standard Care (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (8) | 2 (13)
Hyponatremia (Metabolism and nutrition disorders) | 2 (7) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 2 (5) | 1 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (5) | 1 (2)
Alanine Aminotransferase Increased (Investigations) | 2 (7) | 2 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5) | 1 (4)
Alkaline Phosphatase Increased (Investigations) | 2 (5) | 1 (4) — Alkaline Phosphatase Increased
Dyspnea/Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (3)
Fatigue/Weakness (General disorders) | 2 (8) | 3 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Creatinine Increased (Investigations) | 1 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 1 (4) | 1 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Blood Bilirubin Increased (Investigations) | 1 (7) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GGT Increased (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Slurred speech (Nervous system disorders) | 1 (1) | 0 (0) — Dysarthria
Left arm weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Upper limb weakness
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (4) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Phlebitis (General disorders) | 0 (0) | 1 (1) — Related to gemcitabine
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT04491084/Prot_SAP_000.pdf